CLINICAL TRIAL: NCT06113601
Title: Assessment of Admission to the ICU of Onco-hematological Patients. Income Patterns and Results.
Brief Title: Assessment of Admission to the ICU of Onco-hematological Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital A Coruña (Other)
Responsible Party: Principal Investigator, Elena Cuenca Fito, Principal Investigator, University Hospital A Coruña
Other Study IDs: 23772377
Record Dates: First submitted 2023-07-11; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Hematological Diseases; Critical Illness
MeSH Terms: conditions — Hematologic Diseases; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients admitted to the ICU.
  Interventions: Other: There is no intervention.
- Patients who are not admitted to the ICU.
  Interventions: Other: There is no intervention.

INTERVENTIONS:
Other: There is no intervention. — There is no intervention in the study.

SUMMARY:
Multicenter, observational and prospective study.

DETAILED DESCRIPTION:
The data collection period will include 6 consecutive months, starting from the date of acceptance or conformity of the CEIC. Or, until an adequate sample size is reached that guarantees the statistical relevance of said analysis. All patients will subsequently be followed up 3 months after discharge from the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Solid organ tumor or hematological malignancy,

Exclusion Criteria:

-under 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of solid organ or hematological tumor who are admitted to the hospital and require ICU evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality. | During the 6 months of the study.

IPD SHARING:
Plan to Share IPD: Undecided